CLINICAL TRIAL: NCT01848132
Title: Multicenter Randomized Phase II Study of Treatment With R-CHOP vs Bortezomib-R-CAP for Young Patients With Diffuse Large B-cell Lymphoma With Poor IPI.
Brief Title: Efficacy/Safety Study of R-CHOP vs Bortezomib-R-CAP for Young Patients With Diffuse Large B-cell Lymphoma With Poor IPI.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Grupo Español de Linfomas y Transplante Autólogo de Médula Ósea (Other)
Collaborators: Janssen-Cilag, S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BRCAP-GELTAMO12; 2012-005138-12 (EudraCT Number)
Record Dates: First submitted 2013-05-03; First posted 2013-05-07 (Estimated); Last update posted 2018-09-19 (Actual); Status verified 2018-09

CONDITIONS: Diffuse, Large B-Cell, Lymphoma
Keywords: Lymphoma; Large B-Cell
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Lymphoma | interventions — Bortezomib; Rituximab; Cyclophosphamide; Doxorubicin; Prednisone; Vincristine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- R-CHOP (Active Comparator): 6 cycles every 21 days.
  * Rituximab: intravenous, 375 mg/m2, day 1
  * Cyclophosphamide: intravenous, 750 mg/m2, day 1
  * Doxorubicin: intravenous, 50 mg/m2, day 1
  * Vincristine: intravenous, 1,4 mg/m2, day 1
  * Prednisone: oral, 100 mg, days 1-5
  Interventions: Drug: Rituximab; Drug: Cyclophosphamide; Drug: Doxorubicin; Drug: Prednisone; Drug: Vincristine
- B-R-CAP (Experimental): 6 cycles every 21 days
  * Bortezomib: subcutaneous, 1,3 mg/m2, day 1, 8, 15
  * Rituximab: intravenous, 375 mg/m2, day 1
  * Cyclophosphamide: intravenous, 750 mg/m2, day 1
  * Doxorubicin: intravenous, 50 mg/m2, day 1
  * Prednisone: oral, 100 mg, days 1-5
  Interventions: Drug: Bortezomib; Drug: Rituximab; Drug: Cyclophosphamide; Drug: Doxorubicin; Drug: Prednisone

INTERVENTIONS:
Drug: Bortezomib — Bortezomib: subcutaneous, 1,3 mg/m2, day 1, 8, 15.
  Other Names: Velcade
  Arms: B-R-CAP
Drug: Rituximab — Rituximab: intravenous, 375 mg/m2, day 1
Drug: Cyclophosphamide — Cyclophosphamide: intravenous, 750 mg/m2, day 1
Drug: Doxorubicin — Adriamycin:intravenous, 50 mg/m2, day 1
  Other Names: Adriamycin
Drug: Prednisone — Prednisone: oral, 100 mg, days 1-5
Drug: Vincristine — Vincristine: intravenous, 1,4 mg/m2, day 1
  Arms: R-CHOP

SUMMARY:
Diffuse large B cell lymphoma (DLBCL) is the most common non-Hodgkin's lymphoma, accounting for between 30% and 50% of the patients. Although it is considered a curable disease, still at least 40 % of the patients will fail first line chemotherapy. The International Prognostic Index (IPI) score and the age adjusted IPI (aIPI) has been used since they were published to identify patients with different outcome.

There is not standard therapy for young patients with DLBCL and unfavourable IPI score. The survival of these patients remains poor, with EFS around 40%.

The combination of RCHOP with new drugs is an attractive approach to treat these patients.

The goal is to evaluate the proportion of patients with Event-Free Survival (EFS) after 2 years, with a diagnosis of DLBCL with an aIPI > 1 or an aIPI =1 with increased levels of beta-2-microglobulin (above the Upper Limits of Normal.)

DETAILED DESCRIPTION:
Diffuse large B cell lymphoma (DLBCL) is the most common non-Hodgkin's lymphoma, accounting for between 30% and 50% of the patients. Although it is considered a curable disease, still at least 40 % of the patients will fail first line chemotherapy. The International Prognostic Index (IPI) score and the age adjusted IPI (aIPI) has been used since they were published to identify patients with different outcome.

CHOP chemotherapy administered every 21 days has been for years the standard therapy for advanced DLBCL achieving a long term overall survival (OS) of about 40%. Many studies show that the addition of the monoclonal antibody Rituximab improves the patients survival achieving higher rates of event-free survival in elderly patients with both,favourable and unfavourable IPI score. R-CHOP also improved survival in young patients with favourable IPI score.

There is not standard therapy for young patients with DLBCL and unfavourable IPI score. The survival of these patients remains poor, with EFS around 40%.

The combination of RCHOP with new drugs is an attractive approach to treat these patients.

The investigators propose a phase II randomized clinical trial for young patients with unfavourable IPI score DLBCL using 6 cycles of the combination of subcutaneous Bortezomib with R-CAP (RCHOP without vincristine, to avoid neuropathy) comparing with the standard immunochemotherapy regimen R- CHOP every 21 days.

The goal is to evaluate the proportion of patients with Event-Free Survival (EFS) after 2 years, with a diagnosis of DLBCL with aIPI > 1 or aIPI =1 with increased levels of beta-2-microglobulin (above the Upper Limits of Normal).

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with primary diffuse DLBCL who have never received treatment for this condition.
* Age between 18 and 70 years.
* Age-adjusted IPI (aIPI) higher than 1, or equal 1 with high levels of beta-2-microglobulin (above UNL)
* Cluster of Differentiation 20 (CD20) positive b lymphocytes.
* Eastern Cooperative Oncology Group (ECOG) 0-3.
* More than 12 weeks of life expectancy.
* Signed Informed Consent.
* Nor pregnant women nor breast-feeding women without heterosexual activity during the entire study. Women with heterosexual activity only if they are willing to use two methods of contraceptive. The two contraceptive methods can be, two barrier method or a barrier method combinated with an hormonal contraceptive method to prevent pregnancy, used during the entire study and until 3 months after the study completion.

Exclusion Criteria:

* Pregnant women or in breast-feeding period, or adults in childbearing period not using an effective contraception method.
* Patients with Central Nervous System (CNS) lymphoma.
* Severely impaired renal function (creatinine> 2.5 UNL) or hepatic function impairment (bilirubin or Alanine Amino Transaminase (ALT) / Aspartate Aminotransferase (AST) > 3 UNL), unless it is suspected to be due to the disease.
* Human immunodeficiency virus (HIV) positive patients
* Patient previously treated for the DLBCL
* Positive determination of chronic hepatitis B (defined as positive serology for HBsAg). It will be allowed to enroll patients with hidden or previous hepatitis B (defined as positive antibodies against the core of the hepatitis B virus [HBcAb] and HBsAg negative) if undetectable Hepatitis B Virus (HBV) DNA.
* Positive results for hepatitis C (antibody serology for hepatitis C virus ((HCV)). Patients with HCV positive may only participate if the Polymerase Chain Reaction (PCR) result is negative for HCV RNA.
* History of cardiovascular disease with ventricular ejection fraction < 50%.
* Patients with severe psychiatric conditions that may interfere with their ability to understand the study (including alcoholism or drug addiction).
* Patients with known hypersensitivity to murine proteins or any other components of the study drugs.
* Transformed follicular lymphoma.
* History of other neoplastic malignancy with < 5 year of complete response (except for Squamous Cell Carcinoma of the Skin or cervical Carcinoma in situ).
* Presence of uncontrolled conditions: cardiac, respiratory, neurologic, metabolic etc., not related to lymphoma.
* Uncontrolled hypertension (diastolic blood pressure over 110 mmHg).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2013-10-03 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with Event-Free Survival at 2 years. | During treatment period, there will be assessments every 2 cycles. After end of treatment every 3 month the first year, every 6 months the second year and annually from 3rd to 5th year
  To evaluate the proportion of patients with event-free survival at 2 years in patients diagnosed of DLBCL with aIPI > 1 or aIPI=1 with elevated levels of beta 2-microglobulin (above UNL).
  UNL= Upper Normal Limit.

SECONDARY OUTCOMES:
Event-Free survival at 2 years in the different subtypes of DLBCL | Once the treatment is started, there will be weekly safety visits, visits before each treatment cycle, at day 60 after the sixth cycle and then follow-up visits every three months during the first 2 years and every 6 months until the 5th year
  Event-free survival at 2 years in the different subtypes of DLBCL subgroups: Germinal center B-cell-like (GCB)/non-GCB.
Overall survival at 2 years | Once the treatment is started, there will be weekly safety visits, visits before each treatment cycle, at day 60 after the sixth cycle and then follow-up visits every three months during the first 2 years and every 6 months until the 5th year.
  Overall survival at 2 years in patients diagnosed of DLBCL with aIPI > 1 or aIPI=1 with elevated levels of beta 2-microglobulin (above UNL)
Overall response rate and complete remissions | Once the treatment is started, there will be weekly safety visits, visits before each treatment cycle, at day 60 after the sixth cycle and then follow-up visits every three months during the first 2 years and every 6 months until the 5th year.
  Overall response rate and complete remissions in patients diagnosed of DLBCL with aIPI > 1 or aIPI=1 with elevated levels of beta 2-microglobulin (above UNL).
Toxicity according to the CTC criteria | Once the treatment is started, there will be weekly safety visits, visits before each treatment cycle, at day 60 after the sixth cycle and then follow-up visits every three months during the first 2 years and every 6 months until the 5th year.
  Toxicity according to the Common Toxicity Criteria (CTC) (version 3.0) of the National Cancer Institute (NCI).
To evaluate the predictive value for EFS of interim PET/CT evaluation | Before treatment, after second cycle, after fourth cycle and after treatment completion.
  To evaluate the predictive value for EFS of interim PET/CT evaluation after 2 and 4 cycles of chemotherapy.
  The PET Network group of Grupo Español de Linfomas y Transplante Autólogo de Médula Ósea (GELTAMO), will conduct this blind central review in real-time (qualitative and quantitative, prospective central review of the PET scans performed)
To identify clinical and biological prognostic factors for response and survival. | Once the treatment is started, there will be weekly safety visits, a visit before each treatment cycle, a visit at day 60 after the sixth cycle and then follow-up visits every three months the first 2 years and every 6 months until the 5th year.
  To identify clinical and biological prognostic factors for response and survival.

OTHER OUTCOMES:
Biological project | During recruitment period, after patient randomization.
  * To explore the mutational profile in a selection of these cases by massive sequencing.
  * To analyze the impact of the molecular classification of DLBCL based on immunohistochemistry (IHC) (as Hans algorithms, Choi and Meyer) in the prospective series of the patients of this clinical trial.
  * To explore the effect of the expression of genes, Micro-Ribonucleic Acid (miRNAs) and proteins of interest. Refine the IHC analysis with automatic quantification methods of protein expression.
  * To explore the effect of frequent cytogenetic alterations in DLBCL.

CONTACTS AND LOCATIONS:
Overall Officials: Eva González, MD, Study Chair — Institut Catalá d'Oncología, Hospital Duran i Reynals
Locations (21):
- Spain (21):
  - Hospital Clínico Universitario Lozano Blesa, Zaragoza, Aragon
  - Hospital Son Llàtzer, Palma, Balearic Islands
  - Institut Català d'Oncologia, Hospital Germans Trias i Pujol, Badalona, Barcelona
  - Institut Català d'Oncologia, Hospital Duran i Reynals, L'Hospitalet de Llobregat, Barcelona
  - Hospital Universitario Marqués de Valdecilla, Santander, Cantabria
  - Hospital de Jerez, Jerez de la Frontera, Cádiz
  - Hospital Universitario Fundación Alcorcón, Alcorcón, Madrid
  - Complejo Hospitalario Universitario de Vigo, Vigo, Pontevedra
  - Hospital Universitario Central de Asturias, Oviedo, Principality of Asturias
  - Hospital Clinic i Provincial de Barcelona, Barcelona
  - Hospital Universitari de Girona Doctor Josep Trueta, Girona
  - Hospital Universitario Infanta Leonor, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario La Paz, Madrid
  - Centro Integral Oncológico Clara Campal, Madrid
  - Hospital Universitario de Salamanca, Salamanca
  - Hospital Universitario de Canarias, Santa Cruz de Tenerife
  - Hospital Universitario Virgen del Rocío, Seville
  - Hospital Universitario Doctor Peset, Valencia
  - Hospital Universitari i Politècnic La Fe, Valencia

IPD SHARING:
Plan to Share IPD: No